CLINICAL TRIAL: NCT02511912
Title: Heart Failure (HF) Interatrial Shunt Study 1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was canceled
Sponsor: V-Wave Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HF Study
Record Dates: First submitted 2015-06-30; First posted 2015-07-30 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2016-11

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V-Wave (Experimental): This is a single arm study, all eligible patients will receive the V-Wave implantable shunt.
  The V-Wave device is implanted via standard femoral venous access and inter-atrial septal puncture intervention and is placed through the Fossa Ovalis.
  Interventions: Procedure: V-Wave

INTERVENTIONS:
Procedure: V-Wave — The V-Wave shunt implantation procedure is a standard femoral venous access and inter-atrial septal puncture intervention. The shunt is placed through the Fossa Ovalis.

SUMMARY:
The objective of this study, is to assess the safety and performance of an interatrial shunt when implanted in patients with severe chronic heart failure.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open label, single-arm multi-center study assessing the performance and safety of the V-Wave inter-atrial unidirectional shunt when implanted in chronic heart failure patients with both reduced and preserved ejection fraction.

The V-Wave Interatrial Unidirectional Shunt is designed to enable blood flow in a controlled manner from the left atrium to the right atrium in heart failure patients where clinical sequelae such as symptomatic pulmonary congestion due to high left atrial filling pressure is common.

The objective of this study, is to assess the safety and performance of the V-Wave System when implanted in patients with severe chronic heart failure.

In addition, this study is designed, in-part, to collect a portion of the clinical data needed in support of a US FDA pivotal IDE study application to be submitted at a later date.

Up to 70 subjects with chronic ACC/AHA Stage C, NYHA functional class III or ambulatory class IV heart failure (HF), with reduced or preserved LV ejection fraction, who have a history of hospitalization for worsening HF or elevated ambulatory levels of BNP/NT-proBNP, in the setting of maximally tolerated guideline-directed HF drug and device therapy, will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or non-ischemic cardiomyopathy with either reduced or preserved LV ejection fraction and documented heart failure for at least 6 months
2. ACC/AHA Stage C, NYHA Class III or ambulatory Class IV heart failure,
3. Receiving maximally tolerated medical therapy for heart failure as indicated per ACC/AHA or ESC Heart Failure Guidelines
4. Subject has a minimum of one (1) prior hospital admission within the last 12 months for acute worsening of HF associated with signs/symptoms of congestion
5. Able to perform the 6-minute walk test with a distance ≥150 meters and ≤450 meters.
6. Provide written informed consent for study participation

Exclusion Criteria:

1. Age <18 or >85 years old
2. BMI <18 or >40 kg/m2
3. systolic blood pressure <90 or >160 mmHg
4. Has baseline 2-D echocardiographic evidence of, or history of, unresolved or non- organized intracardiac thrombus
5. Has Pulmonary Hypertension with a pulmonary artery systolic pressure of ≥70 mm/Hg on screening baseline echocardiogram.
6. Significant RV dysfunction defined echocardiographically as TAPSE <12mm or RVFAC ≤30%.
7. Left Ventricular End-Diastolic Diameter (LVEDD) > 8cm
8. Has an Atrial Septal Defect or Patent Foramen Ovale with more than trace shunting on color Doppler or intravenous bubble study or prior surgical or interventional correction of congenital heart disease involving atrial septum including placement of a PFO or ASD closure device
9. Had a Stroke, Transient Ischemic Attack, Systemic or Pulmonary Thromboembolism, or Deep Vein Thrombosis (DVT) within the last 6 months, or any prior stroke with permanent neurologic defect.
10. Has untreated severe stenotic or regurgitant valve lesions, or coronary stenoses which are anticipated to require surgical or percutaneous intervention within 6 months, active valvular vegetations, atrial myxoma, hypertrophic cardiomyopathy with significant resting or provoked subaortic gradient, acute myocarditis, tamponade, or large pericardial effusion, constrictive pericarditis, infiltrative cardiomyopathy (including cardiac sarcoidosis, amyloidosis, and hemochromatosis), or congenital heart disease, as cause of HF.
11. Transseptal procedure is anticipated within 6 months after the V-Wave Shunt implant.
12. Bradycardia with heart rate <45 bpm (unless treated with a permanent pacemaker) or uncontrolled tachyarrhythmias.
13. Intractable HF with resting symptoms despite maximal medical therapy (ACC/AHA HF Stage D).
14. Intolerant to both ACEI and ARB and beta-blocker medical therapy for patients classified as HFrEF (EF ≤40%).
15. Had an acute MI, Acute Coronary Syndrome (ACS), Percutaneous Coronary Intervention (PCI), Rhythm Management system revision, lead extraction, or cardiac or other major surgery within 30 days.
16. Not eligible for emergency open-heart, thoracic or vascular surgery in the event of cardiac perforation or other serious complication during contemplated study device implantation.
17. Has a life expectancy <1 year due to non-cardiovascular illness.
18. Has contraindications to all of the study-related anticoagulation/antiplatelet regimens
19. Has an Estimated Glomerular Filtration Rate <30 ml/min/1.73 m2 by the MDRD method or is receiving dialysis.
20. Hepatic impairment with at least one liver Function Test
21. Severe chronic Pulmonary Disease
22. Active infection requiring systemic antibiotics.

Procedural (final) Exclusion Criteria:

1. Unable to undergo both TEE and ICE.
2. Anatomical anomaly on TEE or ICE
3. Has inadequate vascular access for implantation of shunt.
4. Hemodynamic anomaly or instability at time of FEC

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Freedom from study-related Major Adverse Cardiac and Neurological Events (MACNE) | 6 months
  MACNE is defined as the hierarchical composite of death, stroke, myocardial infarction, systemic embolic event or the requirement for surgical removal of the Study Device.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Mishall, Study Director — V-Wave Ltd
Locations (1):
- V-Wave Ltd., Caesarea Industrial Park (North), Israel

IPD SHARING:
Plan to Share IPD: Undecided